CLINICAL TRIAL: NCT04387903
Title: Surgical Intervention After Pancreaticoduodenectomy: Incidence, Indications, Risk Factors and Outcome
Brief Title: Reoperation After Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hosam Hamed, Lecturer of general surgery, Mansoura University
Other Study IDs: R.20.04.819
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Periampullary Carcinoma; Pancreatic Cancer
Keywords: Pancreaticoduodenectomy, pancreatic fistula, pancreatic cancer, reoperation
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reoperation group: The group of patients who underwent pancreaticduodenectomy for management of periampullary tumors and required surgical reintervention afterwards for management of procedure-related complications as pancreatic fistula, bleeding, abdominal collection, biliary fistula, gastric fistula.
  Interventions: Procedure: Surgical re-interventionafter pancreaticoduodenectomy
- No reoperation group: The group of patients who underwent pancreaticoduodenectomy for management of periampullary tumors and did not require surgical reintervention.
  Interventions: Procedure: Surgical re-interventionafter pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Surgical re-interventionafter pancreaticoduodenectomy — Mandatory surgical management of complications after pancreatico-duodenectomy through peritoneal lavage, draiange, repair of fistula, completion pancreatectomy, control of bleeding, bowel resection, and feeding jejunostomy.

SUMMARY:
The aim of this study is to outline the incidence of early and late reoperation after PD, examine the risk factors for early surgical intervention and its impact on the surgical outcome, hospital stay, diseases recurrence and patient survival, address variable indications for late readmission and reoperation after PD and its impact on patient survival and disease recurrence.

DETAILED DESCRIPTION:
This is a retrospective cohort study of all patients who underwent PD for periampullary tumors in Gastrointestinal Surgical Center (GISC), Mansoura University, Egypt in the period between 2000 and 2018.The exclusion criteria included any patients with locally advanced periampullary tumor, metastases, patients with advanced liver cirrhosis (Child B or C), malnutrition, or coagulopathy.

Patient data were recorded in a prospectively maintained database. Preoperative variables included; age, sex, body mass index, patients' symptoms and signs, laboratory tests, tumor markers and preoperative biliary drainage. Intraoperative variables included; liver status, tumor size, pancreatic duct diameter, texture of the pancreas, operative time, blood loss, pancreatic reconstruction method and blood transfusion. Postoperative variables included postoperative complications, drain amylase, liver function, day to resume oral feeding, postoperative stay, re-exploration, hospital mortality, postoperative pathology, and surgical safety margins.

Data regarding reoperation included incidence, male to female ratio, hospital stay, interval to reoperation, number of explorations, indication of reoperation and surgical management, and postoperative outcome in terms of morbidity and hospital stay. Follow-up was carried out one week postoperatively, 3 months, 6 months and then after one year. The minimum duration of follow up was 2 years. Follow up was done by thorough history taking, clinical examination and abdominal CT in case of suspicious lesions on pelvi-abdominal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent pancreaticoduodenectomy for periampullary malignant lesions in the duration between January 2000 and May 2018

Exclusion Criteria:

* Pancreaticoduodenectomy performed for benign tumors, recurrent malignant tumors, chronic pancreatitis, or inflammatory strictures were excluded from the study.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective cohort study of all patients who underwent PD for periampullary malignant lesions in the duration between January 2000 and May 2018.
  Preoperative assessment was performed by clinical examination and detailed laboratory investigations. Assessment of local extension of the tumor and metastatic work-up was performed by pelvi-abdominal ultrasound (US), triphasic abdominal computerized tomography (CT) with angiographic assessment of the surrounding vessels, bone survey, and chest X-ray. Preoperative endoscopic retrograde cholangiopancreatography (ERCP) for preoperative biliary drainage was performed in selected cases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 2-20 years after surgery
  The duration between surgical intervention to patient death
Tumor recurrence | 2-20 years
  Duration between surgery and recurrence of periampullary tumors based on radiological or endoscopic investigations.

SECONDARY OUTCOMES:
Hospital stay after reoperation | 10-90 days after reoperation
  duration between reoperation surgery to discharge from hospital
Morbidity after reoperation | 10-90 days after reoperation
  complications after reoperation including intr- or extra-luminal hemorrhage, pancreatic or gastric fistula, biliary leakage, thromboembolic diseases, and wound infection
Risk factors for surgical reoperation | Before surgical intervention
  Factors that increase the probability that the patient undergoing pancreaticoduodenectomy would be at higher risk for reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, md, Study Director — Professor of Surgery, Gastrointestinal Surgical Center

IPD SHARING:
Plan to Share IPD: No
The data will be prepared as a research paper and the cohort results will be published in a scientific journal.